CLINICAL TRIAL: NCT01834469
Title: Feasibility Study of the (Intravenously Injected) Indocyanine Green (ICG) Imaging of Tumoral Implants in Patients With Peritoneal Carcinomatosis From Ovarian Carcinoma
Brief Title: Imaging of Peritoneal Carcinomatosis From Ovarian Carcinoma Patients
Acronym: OV-AP-ICG-IV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2083; 2013-000276-15 (Other: Federal Agency for medicine and health products)
Record Dates: First submitted 2013-04-14; First posted 2013-04-18 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-07

CONDITIONS: Ovarian Cancer; Peritoneal Carcinomatosis
Keywords: Ovarian,metastasis
MeSH Terms: conditions — Ovarian Neoplasms; Peritoneal Neoplasms; Krukenberg Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ICG NIR imaging (Other): see Summary and description iv injection of ICG
  Interventions: Drug: iv injection of ICG

INTERVENTIONS:
Drug: iv injection of ICG — An iv injection will be performed for the ovarian cancer patient before the operation.

SUMMARY:
The purpose of this study is to determine if NIF fluorescent imaging is an effective approach to detect the gross ovarian tumoral tissues and peritoneal implants in Ovarian cancer patients.

DETAILED DESCRIPTION:
Primary objective:

Evaluation of the ability of NIR imaging to image and to detect the " viable " gross tumoral mass and/or peritoneal metastatic " implants " in women operated for ovarian carcinoma with peritoneal carcinomatosis after the IV injection of ICG ( which is approved for human use) the day before the operation.

Secondary objective:

Definition of the histological distribution (in the vessels, in the extravascular spaces, in specific cells) of IV injected ICG in the normal and pathological tissues (and, if any is demonstrated pre-operatively, in the nodes of these patients found fluorescent and removed).

however other goals of our project will be will be:

* to confirm that all dissected fluorescent tissue samples are malignant by histopathology.
* to study the histological distribution of ICG in these tumoral tissues.
* to investigate if there is any other florescent tissue in the peritoneal areas which surgeons could not detect any visible tumor implants.
* to distinguish by ICG distribution in between viable tumor tissue from fibrosis and necrosis caused by chemotherapy which is normally difficult to be defined in scars which are routinely removed, but if we could identify the viable tumor tissue by NIF imaging in the operation room, surgeons can avoid dissecting benign scars in the future.

Hopefully ICG will be able to help, firstly, in the scoring of the peritoneal cancer index (PCI) enhancing the detection of small nodules which were undetected by normal visualization allowing a more 'complete' surgical treatment of the disease and secondarily, in the staging of these patients with the potential to upgrade patients from stage I/II to stage III in cases where fluoroscopy would allow to detect unknown minimal peritoneal carcinomatosis.

Methodology:

The day before the operation:

ICG 0.25 mg/kg will be given as an iv injection the day before the operation.

In the operating room:

When the patient will be opened, the surgeons will (under "conventional" video control) search ("in an orderly fashion") and establish "as usual" the presence of "gross" tumoral mass, of metastatic deposits and of "scars" at the level of the peritoneal surfaces. NIR imaging will be acquired during these maneuvers and fluorescent structures and/or foci will be anatomically defined by the surgeons.

The operation will be then continued as usual but each anatomical piece will be controlled "ex vivo" for its fluorescent character or not. All fluorescent foci on these anatomical pieces will be identified as such by a mark and/or by a "suture".

If lymph nodes were suspected to be metastatic (for instance on the basis of the PET-CT with 18F-DG performed before surgery), they will be searched, (optionally controlled in vivo for their visibility using NIR camera)and dissected.

ELIGIBILITY:
Inclusion Criteria:

* Patients (either newly diagnosed, or relapsing) with histo-pathological diagnosis of ovarian carcinoma and peritoneal carcinomatosis who are candidate for "open" surgery, either after neo-adjuvant chemotherapy (80-90% of the cases), or in "first intent".
* Informed consent form signed.

Exclusion Criteria:

* Age less than18 years old.
* Inability to give informed consent.
* History of allergy or hypersensitivity against the investigational product (its active substance or ingredients), to iodine or to shellfish.
* Apparent hyperthyroidism, autonomous thyroid adenoma, unifocal, multifocal or disseminated autonomies of the thyroid gland.
* Documented coronary disease.
* Advanced renal impairment (creatinine > 1,5mg/dl).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Feasibility study of the (intravenously injected) ICG imaging of tumoral implants in patients with peritoneal carcinomatosis from ovarian carcinoma | 1 year
  Evaluation of the feasibility of NIF imaging to detect tumoral implants in patients with peritoneal carcinomatosis from ovarian carcinoma, the efficacy of this approach will be confirmed by histological test of the dissected tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Veys, MD, Principal Investigator — Surgeon in Jules Bordet Institute; Gabriel Liberale, MD, Study Chair — Surgeon in Jules Bordet Institute
Locations (1):
- Jules Bordet Institute, Brussels, Belgium